CLINICAL TRIAL: NCT03235609
Title: Propofol-Ketamine vs. Propofol-Fentanyl for Sedation During Pediatric Diagnostic Gastrointestinal Endoscopy
Brief Title: Sedation During Pediatric Diagnostic Gastrointestinal Endoscopy Gastrointestinal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17100212
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Sedation
MeSH Terms: interventions — Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl (Active Comparator): Group I (FP): will receive 0.5 µg/ kg fentanyl + 2 mg/ kg propofol IV.
  Interventions: Drug: Fentanyl
- Ketamine (Active Comparator): Group II (KP): will receive 0.5 mg/kg ketamine + 2 mg/kg propofol IV.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Fentanyl — fentanyl used with propofol for sedation
  Other Names: Fentanyl Citrate
  Arms: Fentanyl
Drug: Ketamine — ketamine used with propofol for sedation
  Other Names: katalar
  Arms: Ketamine

SUMMARY:
comparison between propofol-fentanyl and propofol-ketamine for sedation in pediatric diagnostic gastrointestinal endoscopy.

DETAILED DESCRIPTION:
It is a prospective double blinded controlled study that will be carried out on 60 pediatric patients undergoing GIT endoscopy; they will be divided into two groups of 30 patients each:- Group I (PF): will receive 0.5 µg/ kg fentanyl + 2 mg/ kg propofol IV. Group II (KF): will receive Ketofol (1 ketamine: 4 propofol) 0.5 mg/kg ketamine + 2 mg/kg propofol IV.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing diagnostic GIT endoscopy
* ASA I-II

Exclusion Criteria:

* Emergency endoscopy
* Respiratory infection and hyperactive airways
* History of serious adverse effects related to anesthetics (e.g. allergic reactions), a family history of reactions to the study drugs
* Morbid obesity, and neuropsychiatric disorders

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-08-16 (Estimated); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
incidence of desaturation | up to 2 days after operation
  when oxygen saturation below 90%

REFERENCES:
- [Background] Michaud L; Francophone Pediatric Hepatology, Gastroenterology, and Nutrition Group. Sedation for diagnostic upper gastrointestinal endoscopy: a survey of the Francophone Pediatric Hepatology, Gastroenterology, and Nutrition Group. Endoscopy. 2005 Feb;37(2):167-70. doi: 10.1055/s-2004-826144. PMID 15692933